CLINICAL TRIAL: NCT01777984
Title: Impact of Visceral Fat on the Pathogenesis of Age-related Macular Degeneration
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rudolf Foundation Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: EK-08-122-0708
Record Dates: First submitted 2011-12-01; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the relationship among the body fat distribution, especially the visceral fat, in patients with age-related macular degeneration in comparison to patients with a normal fundus.

DETAILED DESCRIPTION:
In this study the investigators want to examine the relationship among visceral fat, serum leptin levels, and high-sensitive CRP (hsCRP), Tnf-alpha, Amyloid alpha and Amyloid Beta serum levels in patients with age-related macular degeneration in comparison to patients with a normal fundus.

ELIGIBILITY:
Inclusion Criteria:

* man and women over 18 years old
* filled informed consent
* diagnosis of age-related macular degeneration

Exclusion Criteria:

* inherited retinal disease
* other acquired retinal macular disease
* missing informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with age-related macular degeneration, over 60
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-05 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
visceral fat ratio | 1 day

SECONDARY OUTCOMES:
Leptin, Amyloid, TNF alpha, CRP | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Binder, Principal Investigator — Rudolf Foundation Clinic
Locations (1):
- Rudolf Foundation Clinic, Vienna, Austria, Austria